CLINICAL TRIAL: NCT02730091
Title: A Randomized Open Study of Metronomic Oral Vinorelbine in Combination With Aromatase Inhibitors for the Treatment of Postmenopausal Women With Hormone Receptor Positive,HER2-negative, Advanced Breast Cancer Who Received no Prior Therapy for Advanced Disease
Brief Title: A Open Study of Metronomic Oral Vinorelbine in Combination With Aromatase Inhibitors for the Treatment of Postmenopausal Women With Hormone Receptor Positive,HER2-negative, Advanced Breast Cancer Who Received no Prior Therapy for Advanced Disease
Acronym: VICTORIANE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Collaborators: Pierre Fabre Medicament (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P/2015/253
Record Dates: First submitted 2016-03-25; First posted 2016-04-06 (Estimated); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Letrozole; Anastrozole; Vinorelbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Letrozole or anastrozole (Active Comparator): Letrozole 2,5 mg once a day or anastrozole 1 mg once a day until disease progression, unacceptable toxicity, patient's refusal, consent withdrawal, death, or discontinuation from the study treatment for any other reason.
  Interventions: Drug: Letrozole; Drug: Anastrozole
- Vinorelbine + Anastrozole or letrozole (Experimental): Oral vinorelbine 50 mg (1 soft capsule of 30 mg and 1 soft capsule of 20 mg) three times a week every ( Monday, Wednesday and Friday) before lunch and letrozole 2,5 mg once a day or anastrozole 1 mg once a day until disease progression, unacceptable toxicity, patient's refusal, consent withdrawal, death, or discontinuation from the study treatment for any other reason.
  Interventions: Drug: Letrozole; Drug: Anastrozole; Drug: Vinorelbine

INTERVENTIONS:
Drug: Letrozole — Letrozole 2.5 mg daily
  Other Names: FEMARA
Drug: Anastrozole — anastrozole 1 mg daily
  Other Names: ARIMIDEX
Drug: Vinorelbine — 50 mg three times a week (Monday Wednesday and Friday)
  Other Names: Navelbine
  Arms: Vinorelbine + Anastrozole or letrozole

SUMMARY:
This study is designed to evaluate the clinical effects of the addition of metronomic oral vinorelbine to letrozole and anastrozole. The study will compare the efficacy and tolerability of oral metronomic vinorelbine administered in combination with letrozole or anastrozole, as treatment for hormone receptor-positive advanced or metastatic breast cancer without resistance to Aromatase Inhibitors (AI).

DETAILED DESCRIPTION:
Letrozole and Anastrozole are AI generally used as the first line of therapy for women with HR+ breast cancer.

Furthermore, present hormonal treatments of advanced breast cancer (ABC) or Metastatic breast cancer (MBC) are sub-optimal, as only approximately one half of patients with oestrogen and/or progesterone receptor positive tumours will respond to therapy.

For this patient population, chemotherapy is a valid option, especially after failure or intolerance to hormone therapy. Both combination and sequential single-agent chemotherapy are reasonable options. Based on the available data, sequential monotherapy is recommended as the preferred choice for MBC. Preferred first-line chemotherapy single agents are anthracyclines, taxanes, capecitabine, gemcitabine and vinorelbine.

The development of oral chemotherapy formulations offer numerous benefits to patients, oncologists, oncology nurses, pharmacists and healthcare providers Metronomic therapy (MT) refers to repetitive, low doses of chemotherapy drugs. MT exerts an effect not only on tumor cells, but also on their microenvironment. In particular, the low-dose schedule compromises the repairing process of endothelial cells, leading to an anti-angiogenic effect. A systematic review of the results of phase I, II and III studies suggests that MT is a treatment option for breast cancer patients, has a low toxicity profile, efficacy in most patients and has potentially significant cost-effective advantages for public health.

ELIGIBILITY:
Inclusion Criteria:

* Patient has signed informed consent before any trial related activities and according to local guidelines
* Women with advanced (inoperable loco regionally recurrent or metastatic) breast cancer
* No prior systemic anti-cancer therapy for advanced disease.
* Patient is postmenopausal. Postmenopausal status is defined either by:

  * Prior bilateral oophorectomy
  * Age > 60
  * Age <60 and amenorrhea for 12 or more months (in the absence of chemotherapy, tamoxifen, or ovarian suppression) and/or FSH and estradiol in the postmenopausal range per local normal range
* Patient has a histological and/or cytological confirmed diagnosis of estrogen-receptor positive and/or progesterone receptor positive breast cancer by local laboratory ( determined by >10% positive stained cells for estrogen receptor by IHC on the primary tumor or on metastatic site whichever the value of progesterone receptor).
* Patient has HER2-negative breast cancer defined as a negative in situ hybridization test or an IHC status of 0, 1+ or 2+. If IHC is 2+, a negative in situ hybridization (FISH, CISH, or SISH) test is required by local laboratory testing.
* Patient must have either:

  * Measurable disease, i.e., at least one measurable lesion as per RECIST 1.1 criteria or,
  * At least one lytic bone lesion or . Non measurable disease
* Patient has an Eastern Cooperative Oncology Group (ECOG) performance status <2
* Patient has adequate bone marrow and organ function as defined by the following laboratory values:

  * Absolute neutrophil count ≥ 1.5 × 109/L
  * Platelets ≥ 100 × 109/L
  * Hemoglobin ≥ 8.0 g/dL
  * Normal calcium (corrected for serum albumin)
  * Serum creatinine should be below 2 x ULN
  * In absence of liver metastases, alanine aminotransferase (ALT) and aspartate aminotransferase (AST) should be below 2.5 × ULN. If the patient has liver metastases, ALT and AST should be < 5 × ULN.
  * Total serum bilirubin < ULN; or total bilirubin ≤ 3.0 × ULN with direct bilirubin within normal range of the central laboratory in patients with well documented Gilbert's Syndrome
* Life expectancy > 16 weeks

Exclusion Criteria:

* Patient who received vinorelbine in adjuvant setting.
* Patient with a known hypersensitivity to oral vinorelbine, létrozole, Anastrozole or any of the excipients or others vinca-alcaloïdes. 3. Patient who received any prior anti-cancer therapy (including chemotherapy) for advanced disease with the exception of surgery.

Note:

• Patients who received (neo) adjuvant therapy for breast cancer are eligible. Prior therapy with letrozole or anastrozole in the (neo) adjuvant setting is permitted if the disease free interval is greater than 24 months from the completion of treatment.

* Patient has a concurrent malignancy or malignancy within 5 years of randomization, with the exception of adequately treated, basal or squamous cell carcinoma, non-melanomatous skin cancer or curatively resected cervix cancer.
* Patient with known CNS metastases.
* Patient with impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of the study drugs (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection)
* Patient with a known history of HIV infection (testing not mandatory)
* Patient who any other concurrent severe and/or uncontrolled medical condition that would, in the investigator's judgment, contraindicate patient participation in the clinical study (e.g. chronic pancreatitis, chronic active hepatitis, etc.)
* Patient with active cardiac disease or a history of cardiac dysfunction including any of the following:

History of angina pectoris, symptomatic pericarditis, or myocardial infarction within 6 months prior to study entry History of documented congestive heart failure (New York Heart Association functional classification III-IV) Documented cardiomyopathy

* Patient with peripheral neuropathy>grade 2 CTCAE version 4.0
* Patient who had major surgery within 14 days prior to starting study drug or has not recovered from major side effects
* Patient who concurrently using other antineoplastic agents.
* Patient who has received radiotherapy for palliation ≤ 2 weeks prior to randomization, and who has not recovered to grade 1 or better from related side effects of such therapy (with the exception of alopecia) and/or from whom ≥ 30% of the bone marrow was irradiated.
* Participation in another clinical trial with any investigational drug within 30 days prior to randomization and/or during the study.
* Pregnancy or lactating patients
* Patient with history of surgical resection extended to the stomach or small intestine
* Patient with a severe infection current or recent (within 2 weeks)
* Patient needs long-term oxygen therapy
* Patient with rare hereditary problems of fructose intolerance
* In combination with the vaccine against yellow fever

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2016-02-24 (Actual); Primary Completion 2020-03-23 (Actual); Study Completion 2020-03-23 (Actual)

PRIMARY OUTCOMES:
progression-free survival (PFS) | up to 5 years
  Progression Free Survival is defined as the time from randomization until objective tumor progression or death from any cause if progression did not occur. Subjects will also be considered to have progressed if they have treatment discontinuation with documented evidence of clinical deterioration due to breast cancer. If a patient has not an event, PFS will be censored at the date of the last adequate tumor assessment.

SECONDARY OUTCOMES:
health-related quality of life using HRQoL QLQ-C30 and BR23 | up to 5 years
  using EORTC QLQ-C30 (targeted dimensions: Global Health, physical and Emotional Dimensions, Fatigue and pain) HRQoL will be considered as the first secondary endpoint in order to confirm clinical benefit for the patient since we need more follow up to observe an impact on overall survival (OS).
overall response rate (ORR) | up to 5 years
  ORR and as defined by RECIST 1.1.
clinical benefit rate (CBR) | up to 5 years
  CBR, defined as percentage of patients with complete response (CR), partial response (PR) per RECIST or stable disease (SD) lasting 24 weeks or longer
Safety assessed by NCI CTCAE version 4.0", | up to 5 years
  using NCI CTCAE version 4.0

CONTACTS AND LOCATIONS:
Overall Officials: Erion DOBI, Principal Investigator — Centre Hospitalier Universitaire de Besancon
Locations (1):
- CHU Besançon, Besançon, France